CLINICAL TRIAL: NCT01456156
Title: Phase 2 Study of Postoperative Three-dimensional Conformal Radiation Therapy/Intensive Modulated Radiation Therapy in Hepatocellular Carcinoma: a Single Center Prospective Study
Brief Title: Study of Postoperative 3D-CRT/IMRT in Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Tao Zhang, Principal Investigator, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-019
Record Dates: First submitted 2011-10-12; First posted 2011-10-20 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Hepatocellular Cancer
Keywords: hepatocellular carcinoma; postoperative radiotherapy
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Radiotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hepatectomy plus radiotherapy (Experimental)
  Interventions: Radiation: postoperative radiotherapy

INTERVENTIONS:
Radiation: postoperative radiotherapy — IMRT or 3DCRT, 50-60Gy to the tumor bed
  Other Names: adjuvant radiotherapy

SUMMARY:
Hepatectomy is difficult when the tumor is adjacent to the big vessels of the liver and some patients can not receive radical resection. Such patients have high risk of recurrence. Tumor resection and postoperative radiation is an option for such patients to achieve radical treatment and radiation may reduce local recurrence.

DETAILED DESCRIPTION:
Patients with risk factors of recurrence receive postoperative radiotherapy using intensive modulated radiation therapy (IMRT) or three-dimensional conformal radiation therapy (3DCRT). The clinical target volume includes tumor bed. The dose will be 50-60Gy/25-30f. Overall survival, local-recurrence free survival, disease free survival and toxicity need be observed.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent provided
* 18~75 years old
* patients with histopathological proved hepatocellular carcinoma received hepatectomy and had at least one risk factor of recurrence
* without any lymph node or distant metastasis (any T N0M0)
* liver function: Child-Pugh A or B
* Performance status: Karnofsky (KPS)≥70 or world health organization(WHO) score 0,1
* life expectation>6 months
* no dysfunction of major organs
* no prior radiotherapy
* negative for human immunodeficiency virus syndrome (HIV)
* Considerable to computed tomography(CT) simulation and 3D-CRT or IMRT

Exclusion Criteria:

* malignant tumors of other sits
* combining severe diseases, such as acute myocardial infarction(AMI), arrhythmias, infection
* surgery performed in other hospitals without details
* pregnant woman or woman need to breast feed or woman with positive chorionic gonadotrophin (HCG)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
overall survival | 3 year
  the rate of overall survival for 3 year

SECONDARY OUTCOMES:
local recurrence free survival | 3 years
  the rate of local recurrence free survival for 3 years
disease free survival | 3 years
  the rate of disease free survival for 3 years
Number of Participants with Adverse Events | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Chen B, Wu JX, Cheng SH, Wang LM, Rong WQ, Wu F, Wang SL, Jin J, Liu YP, Song YW, Ren H, Fang H, Tang Y, Li N, Li YX, Wang WH. Phase 2 Study of Adjuvant Radiotherapy Following Narrow-Margin Hepatectomy in Patients With HCC. Hepatology. 2021 Nov;74(5):2595-2604. doi: 10.1002/hep.31993. Epub 2021 Sep 16. PMID 34097307